CLINICAL TRIAL: NCT03377140
Title: Evaluation of the Effects of Hesperidin Supplementation on Hepatic Enzymes, Inflammatory Factors, Lipid Profile, Blood Glucose, Insulin Sensitivity, and Hepatic Steatosis Grade in Patients With Non-alcoholic Fatty Liver Disease
Brief Title: The Effects of Hesperidin on Biochemical Factors and Hepatic Fibrosis in Nonalcoholic Fatty Liver Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Nutrition and Food Technology Institute (Other)
Responsible Party: Principal Investigator, Dr Azita Hekmatdoost, Principal Investigator, National Nutrition and Food Technology Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 6756
Record Dates: First submitted 2017-12-08; First posted 2017-12-19 (Actual); Last update posted 2017-12-19 (Actual); Status verified 2017-04

CONDITIONS: Non Alcoholic Steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Hesperidin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hesperidin (Active Comparator): 2 capsuls of Hesperidin
  Interventions: Dietary Supplement: Hesperidin
- control (Placebo Comparator): 2 capsuls of placebo
  Interventions: Other: control

INTERVENTIONS:
Dietary Supplement: Hesperidin — 2 capsuls
  Arms: Hesperidin
Other: control — 2 capsuls
  Arms: control

SUMMARY:
To study the effects of Hesperidin supplement on lipid profile, liver enzymes, inflammatory factors and hepatic fibrosis in patients with Nonalcoholic Steatohepatitis (NASH), 50 patients who referred to Gastrointestinal (GI) clinic with steatosis grade 2 and 3 will be randomly allocated to receive placebos or 2 capsules Hesperidin for 12 weeks; both groups will be advised to adherence the investigators' diet and exercise program too. At the first and the end of the intervention, lipid profiles, liver enzymes, some inflammatory markers, and liver fibrosis will be assessed and compared between groups.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 to 70 years
* Body Mass Index (BMI) between 25-40
* Sonographic findings compatible with hepatic steatosis (degree 2 or more)

Exclusion Criteria:

* Diabetes
* Taking any kind of antibiotics two weeks before recruitment
* History of alcohol consumption
* pregnancy or lactation
* Professional athletes
* Other liver disease (viral/etc)
* Use of drugs such as calcium channel blockers, high dose synthetic estrogens, methotrexate , amiodarone, steroids, chloroquine, immunosuppressive drugs, lipid-lowering agents, metformin and vitamin E
* A history of Hypertension, Cardiovascular disease, Pulmonary disease, Renal disease & Celiac disease; Cirrhosis
* History of Upper GI surgery / Prior surgical procedures such as jejunoileal or jejunocolic bypass, gastroplasty
* Following program to lose weight in recent 3 mo
* A history of hypothyroidism or Cushing's syndrome

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-02-01 (Estimated); Study Completion 2018-03-20 (Estimated)

PRIMARY OUTCOMES:
liver fibrosis | 12 weeks
  assess by fibroscan

SECONDARY OUTCOMES:
body mass index | 12 weeks
  The body mass index (BMI) or Quetelet index is a value derived from the mass (weight) and height of an individual. The BMI is defined as the body mass divided by the square of the body height, and is universally expressed in units of kg/m2, resulting from mass in kilograms and height in metres.

CONTACTS AND LOCATIONS:
Locations (1):
- National Nutrition and Food Technology Research Institute, Tehran, Iran